CLINICAL TRIAL: NCT04216446
Title: Efficacy of Personalized Mobile-Health Coaching Program During Pregnancy on Maternal Diet, Supplement Use and Physical Activity: a Parallel-Group Randomized Controlled Trial
Brief Title: Mobile Health (m-Health) Coaching Program During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Rozina Nuruddin, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-0757-2504
Record Dates: First submitted 2019-12-20; First posted 2020-01-02 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy
Keywords: m-Health coaching; Pregnancy; Diet; Supplement use; Physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Health Coaching Program during pregnancy (Experimental): Eligible pregnant women would be randomized to intervention or the non-intervention arm after consenting to participate. Participants in the intervention arm will receive free subscription of m-Health program for six months of coaching. The program will provide individualized coaching on diet, supplement use and physical activity. Participants would undergo dietary screening at five points i.e. at baseline and at 6, 12, 18 and 24 weeks follow-up to monitor the improvement (if any) in diet, supplement use and physical activity. Women will receive advice in the form of recommendations after completing the questionnaire. Also, push messages containing tips and recommendations for diet, supplement use and physical activity would be delivered a maximum of three times a week. Furthermore, a subset of participants would undergo objective dietary assessment through biochemical testing of serum folate, serum ferritin, and serum calcium and serum vitamin D at baseline and at end line.
  Interventions: Behavioral: Mobile Health Intervention
- Standard Counseling (No Intervention): For the non-intervention arm, dietary counseling will be provided face to face by the trained research assistant at the baseline and scheduled follow-ups using the AKUH educational leaflet "Diet during Pregnancy" and American College of obstetricians and gynaecologists guidelines for physical activity. Alike intervention group, the non-intervention group will complete an interviewer based paperless screening questionnaire at five points i.e. at baseline and at 6, 12, 18 and 24 weeks follow up. Furthermore, a subset of participants would undergo objective dietary assessment through biochemical testing of serum folate, serum ferritin, and serum calcium and serum vitamin D at baseline and at end line.

INTERVENTIONS:
Behavioral: Mobile Health Intervention — A mobile based application will be developed that will function on android as well as the iPhone operating system. The application will be provided to eligible pregnant women randomized to the intervention group. The dietary, supplement use and physical activity coaching will be provided over the period of 6 months through the application.
  Arms: Mobile Health Coaching Program during pregnancy

SUMMARY:
A parallel-group randomized controlled trial that will evaluate the efficacy of a mobile health (m-Health) program on influencing diet, supplement use and physical activity during pregnancy. Pregnant women will be randomly assigned to the intervention and the non-intervention arm. The intervention arm will receive free of cost m-Health application that will screen on the diet, supplement use and physical activity at enrollment and at 4 follow-ups, each 6 weeks apart. Based on the information provided by women, they will receive personalised recommendations based on an algorithm developed using the World Health Organization's guidelines on nutrition during pregnancy and American College of Obstetricians and Gynaecologists guidelines for physical activity during pregnancy. The non-intervention arm will receive standard face-face counselling. The changes in diet and supplement use of both groups will be assessed using the Dietary Risk Score. Also, biochemical assessment of micronutrients will be carried out on a subset. the change in physical activity will be assessed by the mean duration of reported activity. The secondary outcomes include the evaluation of compliance and usability of the m-Health application. Also, the effect of the m-Health application on maternal, newborn and infant outcomes will be assessed.

DETAILED DESCRIPTION:
A parallel-group randomized controlled trial will be implemented with pregnant women at the antenatal clinics of the Aga Khan University Hospital (AKUH) Karachi. Pregnant women in their first trimester, registered or planning to register at AKUH with access to personal smartphones with internet connection will be considered eligible for the study. For pregnant women in the intervention arm, mobile health application will be provided on their smartphones that will screen their socio-demographic characteristics, diet and supplement use and physical activity habits. Based on the information provided by women, personalized recommendations and a dietary risk score will be generated upon completion of the questionnaire. A similar process will be repeated on 4 follow-ups, each 6 weeks apart after enrollment in the study. Also, push notifications consisting of tips and recommendations will be sent to women a maximum of 3 times a week on dietary, supplement use and physical activity. The women in the non-intervention arm will be provided with standard face-face counselling at similar time points as of intervention group, using the bilingual educational leaflet of the Aga Khan University Hospital "Diet during Pregnancy" and the American College of Obstetricians and Gynaecologists guidelines for physical activity during pregnancy. The primary outcome of the study is improvement in the dietary and supplement use that will be assessed through Dietary Risk Score. A selective subset of participants from both the group will undergo free of cost biochemical assessment micronutrients (serum calcium, vitamin D, iron and folate). The secondary outcomes include assessing the compliance and usability of m-Health application among the pregnant women enrolled in the intervention arm. Other secondary outcomes include evaluating the effect of m-Health coaching on maternal, newborn and infant outcomes among pregnant women in the intervention arm compared to the pregnant women in the non-intervention arm

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women 18 years and above in their first trimester
2. Enrolled at antenatal clinics of The Aga Khan University Hospital, Karachi
3. Pregnant women who have personal smartphones with internet connections.
4. Eligible subjects who consent to participate and agree to remain in the study until the first year of the birth of the baby.

Exclusion Criteria:

1. Pregnant women who have co-morbidity such as cardiovascular disease, diabetes, liver or kidney disease or autoimmune disorder (SLE)
2. Pregnant women who are on dietary control due to co-morbid conditions.
3. Pregnant women who are on platelet aggregates, hypoglycemic or anti-hypertensive drugs.
4. Pregnant women who are unable to read and write due to the language barrier.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Dietary Risk Score (DRS) | 6 months, from enrollment till last follow-up
  Dietary Risk Scores (DRSs) will be calculated based on the consumption of food items from six main food groups and will range from 0-18. Based on the portions and quality of diet, the score for each group will be 0, 1.5 or 3. The total score will be the sum of individual group scores. Higher the aggregate score, poorer the dietary quantity and quality and vice versa. Hence, a score of 18 will indicate a highly inadequate dietary intake; a score of 9 denotes nearly adequate and a score of 0, an adequate diet.
Supplement use Score | 6 months, from enrollment till last follow-up
  Supplement use will be assessed by recording the frequency of consumption of folic acid, iron, calcium and vitamin D in the questionnaire. The frequency will be categorized as daily (7 days a week), often (4-6 days a week) and sometimes (1-3 days a week). Also, a total score ranging from 0-12 will be assigned where each supplement use will be scored 0 for daily, 1.5 for less than daily and 3 for no consumption. The total score will be the sum of each supplement score and will be monitored at each follow-up.
Biochemical Assessment of serum folate at baseline | 1 week of enrollment
  A subset of pregnant women from each group will be selected systematically for the biochemical testing of serum folate at the baseline screening
Biochemical Assessment of serum ferritin at baseline | 1 week of enrollment
  A subset of pregnant women from each group will be selected systematically for the biochemical testing of serum ferritin at the baseline screening
Biochemical Assessment of serum calcium at baseline | 1 week of enrollment
  A subset of pregnant women from each group will be selected systematically for the biochemical testing of serum calcium at the baseline screening
Biochemical Assessment of vitamin D at baseline | 1 week of enrollment
  A subset of pregnant women from each group will be selected systematically for the biochemical testing of vitamin D levels at the baseline screening
Biochemical Assessment of serum folate at endline screening | 24 week of enrollment
  A subset of pregnant women from each group will be selected systematically for the biochemical testing of serum folate at the end line screening.
Biochemical Assessment of serum ferritin at endline screening | 24 week of enrollment
  A subset of pregnant women from each group will be selected systematically for the biochemical testing of serum ferritin at the end line screening.
Biochemical Assessment of serum calcium at endline screening | 24 week of enrollment
  A subset of pregnant women from each group will be selected systematically for the biochemical testing of serum calcium at the end line screening.
Biochemical Assessment of Vitamin D at endline screening | 24 week of enrollment
  A subset of pregnant women from each group will be selected systematically for the biochemical testing of vitamin D levels at the end line screening.
Physical activity | 6 months, from enrollment till last follow-up
  Intensity and duration (minutes) of physical activity will be assessed through the questionnaire at baseline and each follow-up. Household tasks such as cooking, ironing, light physical work, driving and washing dishes will be categorized as mild activities. Brisk walking, gardening, house hold chores such as sweeping, washing, mopping, actively playing with children and carrying loads <20kg will be classified as moderate intensity activities. On the other hand, vigorous intensity activities will include running, fast cycling, aerobics, swimming, sports games or carrying load >20 kg.

SECONDARY OUTCOMES:
Compliance with the intervention | 24 week of enrollment
  Percentage of participants who would complete the six months' program.
Usability of mobile health program | 24 week of enrollment
  Usability of the web-based program will be assessed at the end of the study using a digital evaluation form containing 26 questions with a five response categories Likert-type scale as strongly agree, agree, neutral, disagree and strongly disagree OR always, often, sometimes, rarely and never. it will be assessed under three categories: (i) design and interface, (ii) content and coaching and (iii) perception and personal benefit.
Maternal health outcomes: Pre-eclampsia | Through study completion, average of 1 year
  new onset of hypertension after 20 weeks of gestation along with proteinuria (a spot urine protein/creatinine ratio of ≥30 mg per mmol) and/or evidence of maternal acute kidney injury, liver dysfunction, neurological features, hemolysis or thrombocytopenia, and/or fetal growth restriction.
Maternal health outcomes: Gestational hypertension | Through study completion, average of 1 year
  New onset of hypertension i.e. blood pressure ≥140 mmHg systolic or ≥90 mmHg diastolic at or after 20 weeks' gestation
Maternal health outcomes: Gestational Diabetes | Through study completion, average of 1 year
  Diagnosis made by a single-step 75-g oral glucose tolerance test conducted between 24 and 28 weeks of gestation or at any other time, with one or more of the following results: (1) Fasting plasma glucose 5.1-6.9 mmol/L (92-125 mg/dL); (2) 1-hour post 75-g oral glucose load ≥10 mmol/L (180 mg/dL); (3) 2-hour post 75-g oral glucose load 8.5-11.0 mmol/L (153-199 mg/dL)
Maternal health outcomes: Gestational weight gain during first, second and third trimester | Through study completion, average of 1 year
  Gestational weight gain (GWG) will be determined from weights recorded during the first, second and third trimester. Centiles and z-scores would be assessed using the international gestational weight gain calculator based on the INTERGROWTH-21st standards for gestational weight gain
Newborn birth weight | Through study completion, average of 1 year
  Newborn birth weight in grams adjusted for gestational age at birth will be compared with INTERGROWTH-21st standards.
Newborn length | Through study completion, average of 1 year
  Newborn length in cm adjusted for gestational age at birth will be compared with INTERGROWTH-21st standards.
Preterm birth | Through study completion, average of 1 year
  Preterm births will defined as spontaneous births before completed 37 weeks of gestation.
Infant's Blood Pressure at 1 year | 1 year of infant's age
  Resting blood pressure (BP) would be assessed at 12 month age, after the infant had been calm for >3 min. Mean Systolic and Diastolic BP more than 90th centile appropriate for the height centile and gender will be considered high risk.
Infant's Body Mass Index | 1 year of infant's age
  Infant's weight and length will be assessed at 12 month age.

CONTACTS AND LOCATIONS:
Overall Officials: Rozina Nuruddin, Principal Investigator — Assistant Professor
Locations (1):
- The Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vadsaria K, Nuruddin R, Mohammed N, Azam I, Sayani S. Efficacy of a Personalized mHealth App in Improving Micronutrient Supplement Use Among Pregnant Women in Karachi, Pakistan: Parallel-Group Randomized Controlled Trial. J Med Internet Res. 2025 Apr 9;27:e67166. doi: 10.2196/67166. PMID 40203301
- [Derived] Nuruddin R, Vadsaria K, Mohammed N, Sayani S. The Efficacy of a Personalized mHealth Coaching Program During Pregnancy on Maternal Diet, Supplement Use, and Physical Activity: Protocol for a Parallel-Group Randomized Controlled Trial. JMIR Res Protoc. 2021 Nov 16;10(11):e31611. doi: 10.2196/31611. PMID 34783675